CLINICAL TRIAL: NCT01634776
Title: Behavioral, Genetic, and Epigenetic Implications of Dietary Supplementation With Alpha-linolenic Acid in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Carol Cheatham, PhD, Assistant Professor of Psychology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 09-0358
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Effect of Fatty Acids on Memory Performance of Toddlers
MeSH Terms: interventions — Linseed Oil; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corn oil (Placebo Comparator): 1288 mg/day corn oil
  Interventions: Dietary Supplement: corn oil
- Flaxseed oil (Experimental): 1200 mg/day flaxseed oil
  Interventions: Dietary Supplement: Flaxseed oil

INTERVENTIONS:
Dietary Supplement: Flaxseed oil — Families will be asked to mix the contents of one capsule (1200 mg flaxseed oil or 1288 mg corn oil) into a cup of participants' food, twice a day.
  Arms: Flaxseed oil
Dietary Supplement: corn oil
  Arms: Corn oil

SUMMARY:
Fatty acids or omega-3s are important in the human diet for brain development. Of the three main omega-3s (alpha-linolenic acid: ALA, 18:3n-3; eicosapentaenoic acid: EPA; 20:5n-3; docosahexaenoic acid: DHA, 22:6n-3), DHA and EPA have been studied extensively and have been shown to be important in brain function. Conversely, little is known about the effects of ALA even though the body can make DHA and EPA from it. Because the rate at which ALA makes DHA and EPA is very slow, ALA is not considered an important source of DHA and EPA. However, in the human diet, ALA is more readily available, more easily consumed, and less expensive relative to animal sources of DHA and EPA. So, it is very important that the investigators explore the effects of supplementation with ALA. It is possible that the ALA to DHA and EPA conversion rate can be altered by methylation, an epigenetic form of gene expression and regulation. In the present study, the investigators will examine memory abilities and genetic baselines in 16-month-olds. The investigators will then supplement their food with ALA or control oil for 4 months. At 20 months, the investigators will collect outcome data on memory, fatty acid status, genetic variations, and methylation. The investigators hypothesize that the ALA supplementation will result in an increase in the rate of ALA to DHA and EPA conversion through methylation and genetic variations and subsequently, memory abilities will improve. The data from this study will be used to design a larger R01 grant.

ELIGIBILITY:
Inclusion Criteria:

* 16-month-old toddlers and their natural mothers
* Born fullterm and healthy with no complications
* English as first language

Exclusion Criteria:

* Any toddler with a documented neurological or blood disorder will be excluded.

Ages: 16 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change in declarative memory performance | Baseline, 120 days

SECONDARY OUTCOMES:
Change in fatty acid levels in plasma | Baseline, 120 days
Stability of methylation of promoter region of FADS2 gene | Baseline, 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Carol L Cheatham, Ph.D., Principal Investigator — University of North Carolina, Chapel Hill; Mihai D Niculescu, M.D., Ph.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC at Chapel Hill Nutrition Research Institute, Kannapolis, North Carolina, United States

REFERENCES:
- [Derived] Cheatham CL, Lupu DS, Niculescu MD. Genetic and epigenetic transgenerational implications related to omega-3 fatty acids. Part II: maternal FADS2 rs174575 genotype and DNA methylation predict toddler cognitive performance. Nutr Res. 2015 Nov;35(11):948-55. doi: 10.1016/j.nutres.2015.09.005. Epub 2015 Sep 11. PMID 26455892
- [Derived] Lupu DS, Cheatham CL, Corbin KD, Niculescu MD. Genetic and epigenetic transgenerational implications related to omega-3 fatty acids. Part I: maternal FADS2 genotype and DNA methylation correlate with polyunsaturated fatty acid status in toddlers: an exploratory analysis. Nutr Res. 2015 Nov;35(11):939-47. doi: 10.1016/j.nutres.2015.09.004. Epub 2015 Sep 10. PMID 26439440